CLINICAL TRIAL: NCT05205031
Title: Intravenous Vs. Intraosseous Vascular Access During Out-of-Hospital Cardiac Arrest - a Randomized Clinical Trial
Brief Title: Intravenous Vs. Intraosseous Vascular Access During Out-of-Hospital
Acronym: IVIO
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Lars Wiuff Andersen (Other)
Collaborators: Central Denmark Region (Other); University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Lars Wiuff Andersen, Associate Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 00003
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous (Active Comparator): The intervention will consist of attempts to successfully establish a peripheral intravenous access during the cardiac arrest. The prehospital clinician will be required to attempt the intervention a minimum of two times.
  Interventions: Device: Intravenous
- Intraosseous (Experimental): The intervention will consist of attempts to successfully establish an intraosseous access during the cardiac arrest. The prehospital clinician will be required to attempt the intervention a minimum of two times.
  Interventions: Device: Intraosseous access

INTERVENTIONS:
Device: Intraosseous access — Needle placed in the bone marrow.
  Arms: Intraosseous
Device: Intravenous — Needle placed in a vein.
  Arms: Intravenous

SUMMARY:
The "Intravenous vs. Intraosseous Vascular Access During Out-of-Hospital Cardiac Arrest (IVIO)"-trial is an investigator-initiated, randomized, parallel group, patient and outcome assessor-blinded, superiority trial of intravenous vs. intraosseous vascular access during adult out-of-hospital cardiac arrest. The intraosseous group will be further randomized to humeral vs. tibial access. The trial will be conducted in the Central Denmark Region. The primary outcome will be sustained return of spontaneous circulation, and 762 patients will be included. Key secondary outcomes include survival at 30 days and survival at 30 days with a favorable neurological outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Out-of-hospital cardiac arrest
2. Age ≥ 18 years
3. Indication for intravenous or intraosseous vascular access during cardiac arrest

Exclusion Criteria:

1. Blunt or penetrating traumatic cardiac arrest
2. Prior enrollment in the trial
3. Intravenous or intraosseous vascular access already in place and working when the first trial-participating unit arrives on site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1479 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-05-05 (Actual); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Sustained return of spontaneous circulation | Before or after hospital arrival (up to 2 hours after the cardiac arrest)
  Palpable pulses or other signs of circulation without a need for chest compressions lasting at least 20 minutes

SECONDARY OUTCOMES:
Survival | 30 days after the cardiac arrest
Favorable neurological outcome | 30 days after the cardiac arrest
  Neurological outcome will be assessed with the modified Rankin Scale (mRS) which is a scale from 0 to 6 assessing neurological/functional outcomes after brain damage with higher scores indicating worse neurological/functional outcomes. The scale will will be dichotomized as favorable (mRS 0-3) vs. unfavorable (mRS 4-6).

CONTACTS AND LOCATIONS:
Locations (5):
- Denmark (5):
  - Emergency Medical Services, the North Denmark Region, Aalborg
  - Prehospital Emergency Medical Services, Central Denmark Region, Aarhus N
  - Copenhagen Emergency Medical Services, the Capital Region of Denmark, Ballerup Municipality
  - The Prehospital Center, Region Zealand, Næstved
  - Emergency Medical Services, the Region of Southern Denmark, Vejle

IPD SHARING:
Plan to Share IPD: Yes
Six months after the publication of the last results, all de-identified individual patient data will be made available for data sharing.
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Derived] Vallentin MF, Holmberg MJ, Granfeldt A, Klitgaard TL, Mikkelsen S, Folke F, Christensen HC, Povlsen AL, Petersen AH, Winther S, Frilund LW, Meilandt C, Winther KB, Bach A, Dissing TH, Terkelsen CJ, Christensen S, Rasmussen LK, Mortensen LR, Loldrup ML, Elkmann T, Nielsen AG, Runge C, Klaestrup E, Holm JH, Bak M, Nielsen LR, Pedersen M, Kjaergaard-Andersen G, Hansen PM, Brochner AC, Christensen EF, Nielsen FM, Nissen CG, Bjorn JW, Burholt P, Obling LER, Holle SLD, Russell L, Alstrom H, Hestad S, Fogtmann TH, Hove Buciek JU, Jakobsen K, Krag M, Sandgaard M, Sindberg B, Andersen LW. Intraosseous vs. intravenous access during out-of-hospital cardiac arrest: a Bayesian secondary analysis of a randomised clinical trial. Resuscitation. 2025 Jul;212:110634. doi: 10.1016/j.resuscitation.2025.110634. Epub 2025 May 17. PMID 40348355
- [Derived] Vallentin MF, Granfeldt A, Klitgaard TL, Mikkelsen S, Folke F, Christensen HC, Povlsen AL, Petersen AH, Winther S, Frilund LW, Meilandt C, Holmberg MJ, Winther KB, Bach A, Dissing TH, Terkelsen CJ, Christensen S, Kirkegaard Rasmussen L, Mortensen LR, Loldrup ML, Elkmann T, Nielsen AG, Runge C, Klaestrup E, Holm JH, Bak M, Nielsen LR, Pedersen M, Kjaergaard-Andersen G, Hansen PM, Brochner AC, Christensen EF, Nielsen FM, Nissen CG, Bjorn JW, Burholt P, Obling LER, Holle SLD, Russell L, Alstrom H, Hestad S, Fogtmann TH, Buciek JUH, Jakobsen K, Krag M, Sandgaard M, Sindberg B, Andersen LW. Intraosseous or Intravenous Vascular Access for Out-of-Hospital Cardiac Arrest. N Engl J Med. 2025 Jan 23;392(4):349-360. doi: 10.1056/NEJMoa2407616. Epub 2024 Oct 31. PMID 39480221
- See also: Trial website — https://www.ivio.dk/